CLINICAL TRIAL: NCT02826096
Title: A Brief Version of Biofeedback Therapy for Panic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital, Yun-Lin Branch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201511031RIND
Record Dates: First submitted 2016-07-05; First posted 2016-07-07 (Estimated); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Panic Disorder; Feedback, Psychological
Keywords: Psychiatry; psychological; psychotherapy; randomize; Biofeedback
MeSH Terms: conditions — Panic Disorder | interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- biofeedback group (Experimental): biofeedback therapy
  Interventions: Behavioral: Biofeedback therapy
- medication group (No Intervention): only medication treament

INTERVENTIONS:
Behavioral: Biofeedback therapy — The brief version of biofeedback therapy is conducted by psychologists following the structure way. Biofeedback therapy is six session treatment once a week.
  Arms: biofeedback group

SUMMARY:
The study is to examine the therapeutic effect of a brief version of biofeedback therapy (developed bu the research team) on panic disorder. It is a randomized controlled design. The severity of panic symptoms of two groups of panic patients (reveiving biofeedback therapy or not) were measured before and after the six week duration. Besides, the severity of anxiety, depressive, somatic symptoms, and physiological indexes were recorded.

DETAILED DESCRIPTION:
The purpose of this study is trying to find out whether our newly developed brief version of biofeedback is an effective treatment approach for panic disorder. At the same time, the investigators want to clarify the change of bio- and psycho- indices present through the process. Patient recently experienced panic attacks are recruited in this study. The diagnosis of "Panic Disorder" is made by psychiatrists according to The Diagnostic and Statistical Manual of Mental Disorders(DSM-5) criteria. Subjects are randomly assigned to medication group or biofeedback therapy. The biofeedback therapy is conducted by psychologists following the structure way. Every subject will be measured both the bio and psycho indices on week 0, 3, and 6 under 6-week observation. In the end of the study, the investigators hope to analyze and clarify the treatment effects of our design, and also to exam the meanings of these indices, in order to find out an effective treatment approach.

ELIGIBILITY:
inclusion criteria: The panic disorder cases of the National Taiwan University Hospital Yunlin Branch Psychiatric outpatient department (Huwei, Douliou) have more than one time of panic attack in nearly three months.

exclusion criteria:

1. The age is younger than 20 or older than 70 years.
2. With psychotic symptoms or cognitive dysfunction.
3. A major physical illness (physical illness with fatal risks, such as cancer, myocardial infarction)
4. Unable to read or understand the questionnaire

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-12-21 (Actual); Primary Completion 2021-04-18 (Actual); Study Completion 2021-04-18 (Actual)

PRIMARY OUTCOMES:
Changes from baseline Panic Disorder Severity Scale (PDSS) | week 0, week 3, week 6
  PDSS is a scale rating the severity of panic disorder. It is a 5-point Likert scale with 7 items. The scores range from 0 (lowest level of panic disorder) to 28 (highest level of panic disorder).

SECONDARY OUTCOMES:
Scores of Patient Health Questionnaire-15 (PHQ-15) | week 0, week 3, week 6
  PHQ-15 is a scale rating the severity of somatic distress. It is a 3-point Likert scale with 15 items. The scores range from 0 (lowest level of somatic distress) to 30 (highest level of somatic distress).
Scores of Health Anxiety Questionnaire (HAQ) | week 0, week 3, week 6
  HAQ is a scale rating the severity of health anxiety. It is a 4-point Likert scale with 21 items. The scores range from 0 (lowest level of health anxiety) to 63 (highest level of health anxiety).
Penn State Worry Questionnaire (PSWQ) | week 0, week 3, week 6
  PSWQ is a scale rating the severity of worry. It is 5-point Likert scale with 16 items. The scores range from 1 (lowest level of worry) to 80 (highest level of worry).
Scores of WHOQOL-BREF | week 0, week 3, week 6
  It is a self-report questionnaire measuring health-related quality of life. It is a 4-point Likert scale with 28 items, which belong to 5 domains (the overall, physical, psychological, social and environmental domains). The scores of each domain are usually normalized with 0-20 or 0-100.
Sheehan Function Inventory | week 0, week 3, week 6
  It is a scale rating the function in various dimensions of work, social life, leisure activities, family life and family responsibilities.
Scores of Beck Depression Inventory-II (BDI-II) | week 0, week 3, week 6
  BDI- II is a scale rating the severity of depression. It is a 4-point Likert scale with 21 items. The scores range from 0 (lowest level of depression) to 63 (highest level of depression).
Scores of Beck Anxiety Inventory (BAI) | week 0, week 3, week 6
  BAI is a scale rating the severity of anxiety. It is a 4-point Likert scale with 21 items. The scores range from 0 (lowest level of anxiety) to 63 (highest level of anxiety).
Degree of Change in Physiological Parameters | week 0, week 6
  ProComp5 Infiniti (SA7525) Biofeedback System would be used. Heart rate variability, skin conductance, body temperature and respiratory rate would be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Fu Lin, MD, Principal Investigator — National Taiwan University Hospital, Yun-Lin Branch
Locations (1):
- National Taiwan University Hospital, Douliu, Yun-Lin, Taiwan

IPD SHARING:
Plan to Share IPD: No